CLINICAL TRIAL: NCT03143504
Title: A Longitudinal Investigation of Skin Barrier Development From Birth and the Validation of Early Predictors of Atopic Eczema Risk: the Skin Testing for Atopic Eczema Risk (STAR) Study
Acronym: STAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH19479
Record Dates: First submitted 2017-04-12; First posted 2017-05-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Skin Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin tape-strips (d-squames) containing surface-only corneocytes (dead skin cells).
  Buccal (mouth) swabs. Microbiome swabs from the antecubital fossa (inner elbow joint)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm.: All participants in the same arm.
  Interventions: Diagnostic Test: Skin Testing for Atopic eczema

INTERVENTIONS:
Diagnostic Test: Skin Testing for Atopic eczema — FTIR Spectroscopy. This will involve placing the assessment tool briefly in contact with the baby's skin on the arm and thigh.
  Transepidermal Water Loss. This will involve placing a probe on the baby's skin for approximately 60 seconds on the arm and thigh. The probe measures the rate of water loss from the baby's skin, which indicates how well it acts as a barrier.
  Collection of skin samples. This will involve collecting surface skin samples using small sticky-tape discs to collect only the very top skin cells that are already dead and about to be shed naturally by the body.
  Microbial swab. The researchers will rub the baby's skin gently with a wet sterile swab to collect a sample of the microbes on the baby's skin surface.
  Buccal swab / saliva sample. The researchers will collect a sample of the baby's saliva using a buccal swab. This sample will be used to analyse the baby's genes (DNA) to assess their inherited risk of eczema.

SUMMARY:
Eczema is a chronic disease of the skin that is becoming more common worldwide for reasons unknown. Currently the best indicator that a baby will suffer from eczema is if either or both parents have the condition, although this is not always the case. The goal of this study is to find out if, from birth, the skin of babies who later go on to suffer from eczema develops differently to those who do not. By doing this the research team hope to detect early signs of the disease within the first year of life. Our researchers will ask 150 families from the local Sheffield community to take part in a 1-year study.

To monitor baby skin development, the investigators will carry out 3 simple procedures at the skin surface that pose no risk to the baby. These procedures will be performed on the arm and thigh, at birth, 4 weeks, and 12 months of age. In addition the investigators will ask parents to answer questionnaires and fill out diaries at specific time points throughout the year, to collect information on how they care for their baby's skin. By recording which babies go on to, and do not, develop eczema the investigators hope to: (1) better understand baby skin development from birth, (2) identify if these simple procedures can predict the development of eczema during the first 12 months of life, and (3) investigate environmental effects that may cause disease onset. In a medical era where the prevention of eczema is the long-term goal, it is hoped that this study will provide a new way to identify babies that may go on to develop eczema. This will allow healthcare professionals to offer specific skin care advice from birth, and empower parents to take measured action to help prevent the emergence of eczema in their baby.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the relationship between skin barrier structure/function and skin health in a longitudinal birth cohort. The study (including the purpose and design) has been externally reviewed by a group of peers and was awarded funding by the Leo Foundation.

There is no therapeutic intervention and we will offer no healthcare advice. All participants will be instructed to seek medical care as needed from their normal service provider. As such there are no significant ethical implications.

This study involves a series of harmless procedures to test the properties of the skin in babies and the collection of information on how parents care for their baby's skin over the first 12 months of life. All types of procedures to test the skin are non-invasive and have been used safely in previous clinical studies in babies. Whilst FTIR spectroscopy was used in a previous study conducted by our team in babies (the OBSeRvE study), the investigators will now use a different FTIR instrument. Compared to the benchtop device used for OBSeRvE, the new instrument is better adapted to remote use because of its portability, is safer to use because the measurement head is made of rugged inert materials (diamond and stainless steel) compared to a fragile loop, and the detector is electrically cooled by batteries instead of liquid nitrogen. This device has been tested in humans for safety.

The approach to recruitment of study participants has been informed by the experience of several other clinical studies in babies, including the Barrier Enhancement Eczema Prevention Trial, for which Sheffield has just recently finished recruiting 250 babies. Study recruitment and the skin procedures performed shortly after birth will be led by an experienced Sheffield Teaching Hospitals Research Midwife who is familiar in this clinical environment, and is comfortable with the ethical implications of working with babies and new mothers in the early stages following birth. The Research Midwife will perform the study duties, while remaining sensitive to the needs of the women and babies on the postnatal ward (for example allowing women to breastfeed in peace if requested), and ensuring throughout that maternity service provision will not be adversely affected. The Research Midwife is fully trained in good clinical practice and informed consent. Babies will only be included in the study if the mother's consent is freely provided. Every effort will be made to minimise the burden placed on parents: this means that the researchers will go to the participants to undertake the tests, either at the hospital or at their homes.The researchers will also distribute vouchers to the participants as a "thank you" for their involvement in the study. The voucher amount will be proportionate for their involvement, and is at an appropriate level for the burden of taking part. Taking part is entirely voluntary and the researchers will observe the customs/wishes of the participants. An experienced Research Midwife will lead all hospital assessments, with subsequent follow-up visits being lead by skilled University of Sheffield employed Skin Research Technicians who hold a Sheffield Teaching Hospitals research passport and have undergone a full Disclosure and Barring Services check. All participants will be notified prior to discharge from the maternity ward that the study team conducting home visits consists of both male and female members. If the participant is not happy for a male researcher to conduct a home visit, the researchers will ensure a female member of the team is available as a replacement.

This study includes skin assessments at the participant's home. The research team will complete a lone worker risk assessment and will comply with The University of Sheffield and Sheffield Teaching Hospitals NHS Trust Lone Working guidance. The researchers will issue a study mobile phone for communication during lone working episodes. The researchers have established a set of inclusion and exclusion criteria to ensure that the study is conducted fairly. To ensure that the results are generalizable the researchers have kept the exclusion criteria to a minimum with a geographical restriction centred on the Jessops Wing Maternity Unit established simply for logistical reasons (follow-up sessions being conducted at the participant's homes). The participants will be advised that their data will be held securely, identified only by a unique study number, and that all personal information will be kept strictly confidential. Identifying personal details will be kept only on the study registration form and the Consent form. These documents provide the only link between personal information and the study participant number, and will be kept separately from study data, and stored securely in the STAR study office. Pseudonyms will be used for purposes of transcription and verbatim quotation within any publication. Audio recordings will be destroyed after transcription analysis.

ELIGIBILITY:
Inclusion Criteria:

Mothers 1) ≥18 years old 2) Carrying singleton pregnancies that are booked in to give birth at The Jessop maternity wing (Sheffield Teaching Hospitals NHS Foundation Trust) 3) Live within a 5 mile radius of The University of Sheffield

Babies:

4) Healthy, full-term babies (≥37 weeks gestation) ≤72 hours old

Exclusion Criteria:

Mothers:

1. <18 years old
2. Known to be carrying a baby with a chromosomal abnormality or other syndromic diagnosis
3. Unable to satisfactory give informed consent for participation
4. Multiple pregnancies
5. Live greater than 5 miles from The University of Sheffield

   Babies:
6. Admission to neonatal unit
7. Major congenital malformations or limb defects
8. Illness, social issues or logistical reason that at the discretion of the direct care team, will prevent comfortable trial participation by the family
9. The baby is to be adopted
10. Currently participating in an interventional clinical trial that interferes with the STAR study objectives
11. >72 hours old -

Ages: 37 Weeks to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy, full-term babies (≥37 weeks gestation) ≤72 hours old
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
1) Changes in the molecular structure of the skin from birth (≤72 hours old) to 4 weeks (+2 weeks) and 12 months (±1 month) of age assessed by in-vivo ATR-FTIR spectroscopy | at 4 weeks (+2 weeks), and at 12 months of age (± 1
  As above
Changes in skin barrier function from birth (≤72 hours old) to 4 weeks (+2 weeks) and 12 months (±1 month) of age assessed by TEWL (g/m2/h). | from birth (≤72 hours old) to 4 weeks (+2 weeks) and 12 months (±1 month) of age assessed by TEWL (g/m2/h).
  As above
Changes in desquamatory protease activity (nU μg-1) from birth (≤72 hours old) to 4 weeks (+2 weeks) and 12 months (±1 month) of age determined by ex-vivo laboratory assay. | (≤72 hours old) and at 4 weeks of age (+2 weeks) to predict onset of eczema by 12 months
  As above

SECONDARY OUTCOMES:
Incidence of eczema (UK working party diagnosis) and 'skin rashes' (self-reported) in study participants by 12 months of age. | 12 months
  As above
Diagnostic potential of in-vivo ATR-FTIR spectroscopy, TEWL and desquamatory protease activity measured at birth (≤72 hours old) to predict onset of eczema by 12 months of age using mixed model regression analysis. | 12 months
  As above
Diagnostic potential of in-vivo ATR-FTIR spectroscopy, TEWL and desquamatory protease activity measured at 4 weeks (+2 weeks) to predict onset of eczema by 12 months of age using mixed model regression analysis. | measured at 4 weeks (+2 weeks) to predict onset of eczema by 12 months of age using mixed model regression analysis.
  As above
Incidence of filaggrin loss-of-function mutations within the study population determined by DNA genotyping, and its relationship with skin barrier development / eczema risk by 12 months of age | 12 months
  As above
Capture of information through participant diaries and questionnaires to determine the interaction between the home environment and how parents care for their baby's skin in relation to skin barrier development / eczema risk by 12 months of age. | 12 months
  As above
Capture of parental satisfaction through participant questionnaires on (i) the potential for early diagnosis of skin conditions, (ii) skin care treatments, and (iii) the skin assessments used by this study | 12 months
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Simon G Danby, PhD, BSc, Study Director — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chittock J, Kay L, Brown K, Cooke A, Lavender T, Cork MJ, Danby SG. Association between skin barrier development and early-onset atopic dermatitis: A longitudinal birth cohort study. J Allergy Clin Immunol. 2024 Mar;153(3):732-741.e8. doi: 10.1016/j.jaci.2023.10.017. Epub 2023 Nov 4. PMID 37926123